CLINICAL TRIAL: NCT00002206
Title: A Phase I/II, Double-Blind, Placebo-Controlled Study of the Safety, Tolerance, Pharmacokinetics, and Anti-HIV Activity of 60 Mg Daily Dose of Adefovir Dipivoxil in HIV-Infected Patients Naive to Anti-Retroviral Therapy
Brief Title: A Study of Adefovir Dipivoxil in HIV-Infected Patients Who Have Not Been Treated With Anti-HIV Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 232F; GS-97-420
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-04

CONDITIONS: HIV Infections
Keywords: HIV-1; Adenine; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — adefovir dipivoxil

INTERVENTIONS:
Drug: Adefovir dipivoxil

SUMMARY:
The purpose of this study is to see if it is safe and effective to give adefovir dipivoxil once a day for 4 weeks to HIV-infected patients who never have been treated with anti-HIV medicine. This study also examines how the body processes adefovir dipivoxil.

DETAILED DESCRIPTION:
This a double-blind, placebo-controlled, randomized Phase I/II study of the safety, tolerance, pharmacokinetics, and anti-HIV activity of adefovir dipivoxil in HIV-infected patients naive to antiretroviral therapy. Patients are randomized to receive a single daily dose of adefovir dipivoxil or matching placebo tablet for 4 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection, as indicated by a history of seropositivity for HIV-1 infection (ELISA confirmed with Western blot).
* Peripheral blood CD4 cell count greater than or equal to 150 cells/mm3 on at least 1 measurement within 28 days prior to enrollment.
* Plasma HIV-1 RNA greater than or equal to 5,000 copies/ml within 28 days of study entry.
* A minimum life expectancy of 12 months.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* Active, serious infections (other than HIV infection) requiring parenteral antibiotic therapy. Patients should be considered recovered from such infectious episodes when at least 2 weeks have elapsed following the cessation of parenteral antibiotic therapy.
* Evidence of a gastrointestinal malabsorption syndrome or inability to receive an orally-administered medication.
* A malignancy other than cutaneous Kaposi's sarcoma (KS). (NOTE:
* Patients with biopsy-confirmed KS are eligible, but must not have received any systemic therapy (including chemotherapy) for KS within 4 weeks prior to study entry.

  1. Antiretroviral therapy, including nucleoside analogues, nonnucleoside reverse transcriptase inhibitors, protease inhibitors, or investigational antiretroviral agents (antiretroviral therapy may be started after completion of the Day 35 follow-up visit).
* Interferon (alpha, beta, or gamma) or interleukin (e.g., IL-2).
* Aminoglycoside antibiotics, amphotericin B, cidofovir, diuretics, foscarnet, ganciclovir, itraconazole, fluconazole, ketoconazole (topical allowed), isoniazid, rifampin, rifabutin, clarithromycin, azithromycin, chemotherapeutic agents (systemic), systemic corticosteroids, other agents with significant nephrotoxic potential, other agents that inhibit or compete for elimination via active renal tubular secretion (e.g., probenecid), and other investigational agents.

  1. Treatment with any HIV protease inhibitor.
* Treatment for more than a total of 2 weeks with any nucleoside or nonnucleoside reverse transcriptase inhibitor antiretroviral agent.
* Ongoing treatment with interferon (alpha, beta, or gamma), interleukins or other immunomodulatory agents, systemic corticosteroids, or any investigational agents except on sponsor's approval within 1 month prior to study entry.

Evidence of active substance abuse (including alcohol), as determined by the investigator, that would preclude adequate compliance with the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Anderson Clinical Research, Washington D.C., District of Columbia
  - Johns Hopkins Univ Clinical Pharmacology, Baltimore, Maryland
  - Anderson Clinical Research, New York, New York
  - Anderson Clinical Research, Philadelphia, Pennsylvania
  - Anderson Clinical Research / Inc, Pittsburgh, Pennsylvania